CLINICAL TRIAL: NCT06897852
Title: Accuracy of Photogrammetric Three-Dimensional Facial Models Reconstruction Compared With Direct Anthropometry
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Assem Hammas, Principal Investigator, Al-Azhar University
Other Study IDs: AlAzharU-AZUD
Record Dates: First submitted 2023-07-17; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Dental Malocclusion; Diagnosis; Facial Asymmetry
Keywords: facial scanning; photogrammetry; facial anthropometry
MeSH Terms: conditions — Malocclusion; Disease; Facial Asymmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Direct facial anthropometry group
- first photogrammetric software group
- second photogrammetric software group

SUMMARY:
Accuracy of Two Different Photogrammetric Software for Three Dimensional Facial Model Reconstructions Compared with Direct Facial Anthropometry.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 or older

Exclusion Criteria:

* Presence of:

  1. Extensive facial hair (beards).
  2. Significant facial defects.
  3. Surgical scars.
  4. Neuromuscular disorders that may hinder stability of head during image acquisition.
  5. Accessories that could interfere with image acquisition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be carried out on fifty volunteers, selected from outpatient clinic at Department of Orthodontics, Faculty of Dental Medicine, Al-Azhar University, Assiut branch; aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of Photogrammetry in Generating 3D Facial Models - Linear Measurements | Baseline (procedure)
  * A 3D model was generated for each volunteer using photogrammetry software. Anthropometric linear measurements was taken using a digital caliper, and photogrammetric linear measurements was extracted from the 3D model.
  * Two LEGO® blocks with uniform dimensions were attached to the participants' faces to scale the 3D model to actual metric dimensions.
  Unit of Measure: millimeters(mm)
Accuracy of Photogrammetry in Generating 3D Facial Models - Angular Measurements | Baseline (procedure)
  * This outcome measure focuses on the accuracy of photogrammetry in capturing and reproducing angular measurements of facial features.
  * Volunteers' 3D facial models were generated using photogrammetry software from multiple photos.
  * Two LEGO® blocks with uniform dimensions were attached to the forehead and cheek for scaling and reference. Angular measurements, based on these blocks, were extracted from the 3D model. The measurements were compared to validate the method's precision in reproducing angular dimensions.
  Unit of Measure: Degrees (°)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Al-Azhar University, Asyut, Egypt

REFERENCES:
- [Background] Bradley E, Shelton A, Hodge T, Morris D, Bekker H, Fletcher S, Barber S. Patient-reported experience and outcomes from orthodontic treatment. J Orthod. 2020 Jun;47(2):107-115. doi: 10.1177/1465312520904377. Epub 2020 Feb 29. PMID 32116083
- [Background] Sarver DM. Interactions of hard tissues, soft tissues, and growth over time, and their impact on orthodontic diagnosis and treatment planning. Am J Orthod Dentofacial Orthop. 2015 Sep;148(3):380-6. doi: 10.1016/j.ajodo.2015.04.030. PMID 26321335
- [Background] Mohan A, Sivakumar A, Nalabothu P. Evaluation of accuracy and reliability of OneCeph digital cephalometric analysis in comparison with manual cephalometric analysis-a cross-sectional study. BDJ Open. 2021 Jun 17;7(1):22. doi: 10.1038/s41405-021-00077-2. PMID 34140466
- [Background] Kamburoglu K. Use of dentomaxillofacial cone beam computed tomography in dentistry. World J Radiol. 2015 Jun 28;7(6):128-30. doi: 10.4329/wjr.v7.i6.128. PMID 26120381
- [Background] Jain S, Choudhary K, Nagi R, Shukla S, Kaur N, Grover D. New evolution of cone-beam computed tomography in dentistry: Combining digital technologies. Imaging Sci Dent. 2019 Sep;49(3):179-190. doi: 10.5624/isd.2019.49.3.179. Epub 2019 Sep 24. PMID 31583200
- [Background] Mao WY, Lei J, Lim LZ, Gao Y, Tyndall DA, Fu K. Comparison of radiographical characteristics and diagnostic accuracy of intraosseous jaw lesions on panoramic radiographs and CBCT. Dentomaxillofac Radiol. 2021 Feb 1;50(2):20200165. doi: 10.1259/dmfr.20200165. Epub 2020 Sep 17. PMID 32941743
- [Background] Struck R, Cordoni S, Aliotta S, Perez-Pachon L, Groning F. Application of Photogrammetry in Biomedical Science. Adv Exp Med Biol. 2019;1120:121-130. doi: 10.1007/978-3-030-06070-1_10. PMID 30919299
- [Background] Heike CL, Upson K, Stuhaug E, Weinberg SM. 3D digital stereophotogrammetry: a practical guide to facial image acquisition. Head Face Med. 2010 Jul 28;6:18. doi: 10.1186/1746-160X-6-18. PMID 20667081
- [Background] Erten O, Yilmaz BN. Three-Dimensional Imaging in Orthodontics. Turk J Orthod. 2018 Sep;31(3):86-94. doi: 10.5152/TurkJOrthod.2018.17041. Epub 2018 Apr 11. PMID 30206567
- [Background] D'Ettorre G, Farronato M, Candida E, Quinzi V, Grippaudo C. A comparison between stereophotogrammetry and smartphone structured light technology for three-dimensional face scanning. Angle Orthod. 2022 May 1;92(3):358-363. doi: 10.2319/040921-290.1. PMID 35015071
- [Background] 12- Arapovic-Savic M, Savic M, Umicevic-Davidovic M, Arbutina A, Nedeljkovic N, Glisic B. A novel method of photogrammetry measurements of study models in orthodontics. Srpski arhiv za celokupno lekarstvo. 2019;147(1):10-6.
- [Background] Gupta A. On imaging modalities for cephalometric analysis: a review. Multimedia Tools and Applications. 2023 Mar 21:1-22.